CLINICAL TRIAL: NCT02312804
Title: A Phase Ib Study Evaluating BGJ398 in Combination With Chemotherapeutic Regimen in Patients With Stage IV, Recurrent or Persistent Carcinoma of The Cervix and Other Solid Tumors
Brief Title: Ph Ib/BGJ398/Cervix and Other Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug not available.
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Steven Weitman, Clinical Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTMS 14-2006
Record Dates: First submitted 2014-10-01; First posted 2014-12-09 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Cancer of Cervix; Tumors
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms | interventions — infigratinib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose Escalation (Experimental): To determine the MTD/RP2D of BGJ398 when combined with carboplatin and paclitaxel in subjects with locally advanced for metastatic solid tumors.
  Interventions: Drug: BGJ398; Drug: Carboplatin; Drug: Paclitaxel
- Expansion Cervical Cancer (Experimental): To assess the anti-tumor effect of BGJ398 when combined with carboplatin and paclitaxel in cervix cancer.
  Interventions: Drug: BGJ398; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: BGJ398 — BGJ398 will be administered orally once daily on each day of the 21 day cycle.
  Other Names: BGJ 398
Drug: Carboplatin — Carboplatin will be administered in combination with paclitaxel intravenously on the first day of each 21-day cycle.
  Other Names: Paraplatin
Drug: Paclitaxel — Paclitaxel will be administered in combination with carboplatin intravenously on the first day of each 21-day cycle.
  Other Names: Taxol

SUMMARY:
This study will be conducted using 3+3 design and includes, a dose escalation part to define the MTDfRP2D for the combination of BGJ398 and carboplatin/paclitaxel, and a dose expansion part to treat another 12 patients (only cervix cancer) to further evaluate safety of this combination. Safety, tolerability and MTD will be determined in the dose escalation part of the study. The dose expansion will additionally investigate preliminary anti-tumor efficacy in cervical cancer. The dosing cycle is 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age >18 years at the time of informed consent
* Histologically/cytologically confirmed locally advanced or metastatic solid tumors for which no curable therapy exists. In dose expansion part of this study, only patients with stage IV or recurrent/persistent cervical cancer will be enrolled. Confirmation of FGF/FGFR aberration is not required.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Adequate marrow function as defined below:

absolute neutrophil count ≥ 1.5 x 10 9/L platelets ≥ 100,000 x 10 9/L hemoglobin ≥ 9.0 g/dL Adequate liver function as evidenced by bilirubin <1.5 times the upper limit of normal (ULN); alanine aminotransferase (AL T) and aspartate aminotransferase (AST) <3 times the ULN

* Evidence of measurable or evaluable disease, as determined by RECIST v 1.1
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: has not undergone a hysterectomy or bilateral oophorectomy, or has not been naturally postmenopausal for at least 12 consecutive months (Le., has had menses at any time in the preceding 12 consecutive months). Oral contraceptives (OC), injected or implanted hormonal methods are not allowed as the sole method of contraception because BGJ398 has not been characterized with respect to its potential to interfere with PK and/or the effectiveness of OCs.
* It is preferred that archival tumor sample is available for molecular testing, if not available, a newly obtained tumor biopsy may be submitted instead (not mandatory)

Exclusion Criteria:

* For patients enrolled in dose escalation, any number of prior treatments allowed. For patients enrolled in dose expansion, no prior chemotherapy is allowed (previous single agent cisplatin concurrent with radiotherapy is accepted).
* No prior therapy with paclitaxel, BGJ398 or other FGFR targeting agents.
* Preexisting> grade 2 peripheral neuropathy
* Patients with brain metastases are allowed provided that they are clinically stable for a period of 30 days prior to study entry and there is not a requirement for steroids or anti epileptics.
* History of pancreatitis in last 6 months prior to enrollment.
* History and/or current evidence of endocrine alterations of calcium/phosphate homeostasis, e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis, or patients with other phosphate regulating abnormalities. Because hyperphosphatemia is a frequent occurrence with BGJ398 treatment, pretreatment and concurrent treatment with phosphate regulating agents is allowed.
* Current evidence of corneal or retinal disorder/ keratopathy such as bullous/ band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjunctivits, etc
* Since BGJ398 is a likely inhibitor of CYP3A4, patients who are currently receiving treatment with agents that are known sting inducers or inhibitors CYP3A4 are not allowed
* Treatment with any of the following anti-cancer therapies prior to the first dose of the of BGJ398 within the stated timeframes: intravenous chemotherapy within a period of 4 weeks ( 6 weeks for nitrosourea, mitomycin-C), biological therapy (e,g. antibodies) within a period of time that is ~ 5 t1/2 or less than 4 weeks, whichever is shorter, prior to starting study drug, any other investigational agents within a period of time that is < 5 tl/2 or 4 weeks (whichever is shortest) prior to starting study drug, wide field radiotherapy < 4 weeks or limited field radiation for palliation < 2 weeks prior to starting study drug.
* Use of medications that increase serum levels of phosphorus and/or calcium.
* History of cardiac disease (Congestive heart failure NYHA grade> 2, LVEF < 50% as determined by MUGA scan or ECHO, history of clinically significant ventricular arrhythmias, unstable angina pectoriS or acute myocardial infarction <6 months prior to starting study drug, QTcF > 450 msec)
* Pregnant or nursing (lactating) women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) based on toxicity analysis. | approximately 12 months
  Toxicity will be monitored according to NCI Common Toxicity Criteria for Adverse Events (CTCAE), Version 4.0.

SECONDARY OUTCOMES:
Time vs. concentration profile of BGJ398 | At Cycle 1 Day 1 and Cycle 2 Day 1
  Plasma concentration versus time profiles. Plasma PK parameters will be used to characterize the PK profiles of BGJ398 when combined with certain chemotherapies.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Weitman, MD, Principal Investigator — Clinical Investigator